CLINICAL TRIAL: NCT02196259
Title: Anesthesia and Brain Functional Connectivity: An Analysis of fMRI Changes in Chronic Pain and Refractory Depression
Brief Title: Anesthesia and Functional Connectivity: An Analysis of fMRI Changes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding cessation.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Scott Peltier, Associate Research Scientist, Biomedical Engineering, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: U028860-MICHR-Pilot
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-03

CONDITIONS: Changes in Brain Network Connectivity
Keywords: Pre-Post
MeSH Terms: interventions — Anesthetics, Dissociative; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Initial MRI (Experimental): The subject will receive intravenous ketamine anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Interventions: Drug: Anesthetics, Dissociative
- Initial hospital (Experimental): The subject will receive intravenous ketamine anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Interventions: Drug: Anesthetics, Dissociative
- Depression MRI (Experimental): The subject will receive intravenous ketamine anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Interventions: Drug: Anesthetics, Dissociative

INTERVENTIONS:
Drug: Anesthetics, Dissociative — The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Other Names: Ketamine

SUMMARY:
Functional connectivity is defined as a correlation in neural activity between distinct regions of the brain. Several recent studies have demonstrated areas of low-frequency functional connectivity inherent to brain tissue at rest. These oscillations can be measured using functional magnetic resonance imaging (fMRI) and appear to be synchronized between related areas of the brain.

To date, no investigators have examined the effects of low-dose anesthesia on functional connectivity. This study will image the human brain under conditions of rest, and low-dose anesthetic induced sedation. Quality of the acquired signals will be evaluated and functional networks in the brain will be examined. Of interest is whether administration of a low-dose anesthetic disrupts functional connectivity in the brain, and whether a disruption of functional connectivity is responsible for the reported analgesic and antidepressant effects of a anesthetic.

Participation in the study includes four visits: an in-person interview, an initial fMRI scan, the anesthesia infusion, and a second fMRI scan. There is an optional follow-up fMRI scan one week post infusion.

DETAILED DESCRIPTION:
Background:

A phencyclidine derivative developed by Parke-Davis represented an attempt to mimic phencyclidine anesthesia without inducing the severe psychomimetic reactions of its parent compound. Initial reports were promising and received great enthusiasm. At high doses, the drug was found to provide profound analgesia whilst preserving airway reflexes. It induced reliable amnesia, yet could be delivered as a simple injection. It was claimed at the time that this anesthetic heralded a new phase in the history of anesthesia. Today, over 40 years since the anesthetic was introduced at Michigan, there has been a resurgence of interest in this old drug. A growing number of investigators are studying the effects of anesthesia on human subjects. There is currently tremendous interest in anesthesia as an opioid sparing agent, a model for schizophrenia, an antidepressant, and as an N-Methyl D-Aspartate (NMDA) antagonist in complex regional pain syndromes.

Functional connectivity is a measure of low-frequency oscillations (<0.08 Hz) that are inherent to brain tissue at rest. These oscillations are measured on fMRI, and appear to be synchronized between related areas of the brain. Although research in this area is still in its infancy, studies of the motor, auditory, visual, and sensorimotor systems, have shown that functionally related areas of the brain produce correlated low-frequency oscillations. This fascinating finding raises the possibility of a new approach to studying brain function as well as a potential tool for the diagnosis of disease. Recent fMRI studies of the precentral gyrus have demonstrated the ability of functional connectivity studies to differentiate healthy volunteers from patients with multiple sclerosis. Additional research is ongoing to determine whether functional connectivity will prove useful in the diagnosis of early Alzheimer's disease.

Recent research in functional connectivity has identified regions in the brain active at rest. These regions are often referred to at the "Default-mode network" (DMN). Activity in the DMN is increased in the brain at rest and decreased when a subject concentrates on a mental task. The first fMRI study examining functional connectivity in chronic pain patients was published in a recent issue of the Journal of Neuroscience. In this study abnormal patterns of functional connectivity were seen in chronic pain patients. Specifically, a dysfunction in down-regulating the DMN was seen. The chronic pain patients did not deactivate the medial prefrontal cortex, amygdala, or posterior cingulate cortex to the same degree as healthy controls.

The only fMRI study examining functional connectivity in major depression was published in September of 2007. This study also noted a dysfunction in the DMN. Depressed subjects were found to have increased network functional connectivity in the subgenual cingulate cortex, thalamus, orbitofrontal cortex, and the precuneus. Notably, the subgenual cingulate cortex is the location of a recent clinical trial suggesting that deep brain stimulation to this region may ameliorate symptoms of patients with severe refractory depression.

Interest in anesthesia for the treatment of chronic pain and depression has grown in recent years. Although there have been no randomized trials of low-dose anesthesia in chronic pain patients, the evidence currently available indicates it is most effective in the treatment of allodynia, hyperalgesia, and hyperpathia. For depression, there has been one randomized, placebo-controlled, double blinded crossover study. In the depression trial, robust and rapid antidepressant effects were found to result from a single intravenous dose of anesthesia and last for at least a week.

Objective:

To examine functional connectivity in the human brain both at rest and after anesthetic sedation using functional magnetic resonance imaging (fMRI).

Specific Aims/Hypotheses:

1. Measure the degree of functional connectivity in three study groups (healthy volunteers, chronic back pain, and refractory depression).
2. Analyze for differences in baseline functional connectivity.
3. Measure changes in functional connectivity after IV low-dose anesthetic sedation.
4. Document study group differences in anesthetic response.
5. Measure for any correlation between fMRI changes and therapeutic effects.

Study Protocol:

Participation in this study includes four main visits and an optional follow-up visit. The first visit is a baseline interview session to assess participant eligibility using a structured interview. The second visit is an initial fMRI scan at the fMRI center. The third visit is the anesthetic infusion at the hospital; management of any adverse events during the infusion will be monitored by the Post Anesthesia Care Unit ( PACU) personnel. The fourth visit is a follow-up fMRI scan at the fMRI center. There is an optional one week follow-up visit at the fMRI center for a final fMRI scan.

fMRI Statistical Analysis: The imaging experiments and analysis of subject-specific data will lead to maps corresponding to separate measures: resting state functional connectivity maps, and measures of cerebral blood flow (CBF). Final inferences will be made at the voxel level and for anatomically specific regions-of-interest (ROIs). The voxel-based analysis will be performed through the generation of summary images referred to as statistical parametric maps (SPMs) representing before-infusion vs. after-infusion, and, as data in the two patient groups become available, two-way ANOVA results of ketamine infusion state and patient diagnosis (chronic pain or refractory depression). The ROI-based analysis will be driven by the a priori selected fronto-limbic regions of interest generated in the self-reflection task, and by the anatomical nodes in the default mode network given in the literature.

ELIGIBILITY:
Control Group:

Inclusion Criteria:

(4) Ability to tolerate small, enclosed spaces without anxiety; (6) English fluency.

Exclusion Criteria:

* Pregnant or trying to become pregnant.
* history of serious head injury;
* possibility of ferrous metals within the body, e. g. aneurysm clips, retained particles; or metal that would impair the magnetic resonance (MR) signal, e.g., some dental hardware;
* Smoking usage > 10 cigarettes per day
* Daily intake of caffeine exceeds 2 cups of coffee per day
* Unstable cardiac problems (e.g. severe or poorly treated hypertension, unstable arrhythmia, etc.) or concurrent medications for which anesthesia would be contraindicated
* Patients with a current general medical illness that is life threatening or inadequately treated will be excluded: moderate-to-severe chronic pain, evidence of fracture or malignancy, inflammatory joint disease, severe physical impairment (e.g., bilateral amputation, blindness), morbid obesity, autoimmune/inflammatory diseases, cardiopulmonary disorders (i.e., angina, congestive heart failure, COPD), chronic renal insufficiency, uncontrolled endocrine or allergic disorders (i.e., hyper-/hypothyroidism, diabetes, allergic rhinitis), malignancy.
* Taking any medication, prescription or non-prescription, with psychotropic effects.
* History of psychiatric or neurological illness; History of substance abuse or dependence Positive urine toxicology screen.

Refractory Depression Group:

* Meets all above control group screening criteria except history of psychiatric illness and prescription medication usage
* Included subjects will have a Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) diagnosis of major depressive disorder, recurrent or chronic, moderate-to-severe, without psychotic features, with medication resistance, accepted with agreement by two different psychiatrists. For this study, treatment resistance is defined as ≥2 failed adequate antidepressant trials.
* Patients with a DSM-IV diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder will be excluded. Any history of antidepressant- or substance- induced hypomania or mania will be excluded.
* Subjects will be free of comorbid substance abuse or dependence for at least 3 months, with a negative urine toxicology screen.
* No current suicide plan or intent.
* Comorbid Axis I anxiety disorder diagnoses will be permitted if they do not require current treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Peltier, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - fMRI Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Lowe MJ, Mock BJ, Sorenson JA. Functional connectivity in single and multislice echoplanar imaging using resting-state fluctuations. Neuroimage. 1998 Feb;7(2):119-32. doi: 10.1006/nimg.1997.0315. PMID 9558644
- [Background] Cordes D, Haughton VM, Arfanakis K, Wendt GJ, Turski PA, Moritz CH, Quigley MA, Meyerand ME. Mapping functionally related regions of brain with functional connectivity MR imaging. AJNR Am J Neuroradiol. 2000 Oct;21(9):1636-44. PMID 11039342
- [Background] Lowe MJ, Phillips MD, Lurito JT, Mattson D, Dzemidzic M, Mathews VP. Multiple sclerosis: low-frequency temporal blood oxygen level-dependent fluctuations indicate reduced functional connectivity initial results. Radiology. 2002 Jul;224(1):184-92. doi: 10.1148/radiol.2241011005. PMID 12091681
- [Background] Baliki MN, Geha PY, Apkarian AV, Chialvo DR. Beyond feeling: chronic pain hurts the brain, disrupting the default-mode network dynamics. J Neurosci. 2008 Feb 6;28(6):1398-403. doi: 10.1523/JNEUROSCI.4123-07.2008. PMID 18256259
- [Background] Greicius MD, Flores BH, Menon V, Glover GH, Solvason HB, Kenna H, Reiss AL, Schatzberg AF. Resting-state functional connectivity in major depression: abnormally increased contributions from subgenual cingulate cortex and thalamus. Biol Psychiatry. 2007 Sep 1;62(5):429-37. doi: 10.1016/j.biopsych.2006.09.020. Epub 2007 Jan 8. PMID 17210143
- [Background] Mayberg HS, Lozano AM, Voon V, McNeely HE, Seminowicz D, Hamani C, Schwalb JM, Kennedy SH. Deep brain stimulation for treatment-resistant depression. Neuron. 2005 Mar 3;45(5):651-60. doi: 10.1016/j.neuron.2005.02.014. PMID 15748841
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Woods RP, Grafton ST, Holmes CJ, Cherry SR, Mazziotta JC. Automated image registration: I. General methods and intrasubject, intramodality validation. J Comput Assist Tomogr. 1998 Jan-Feb;22(1):139-52. doi: 10.1097/00004728-199801000-00027. PMID 9448779
- [Background] Tzourio-Mazoyer N, Landeau B, Papathanassiou D, Crivello F, Etard O, Delcroix N, Mazoyer B, Joliot M. Automated anatomical labeling of activations in SPM using a macroscopic anatomical parcellation of the MNI MRI single-subject brain. Neuroimage. 2002 Jan;15(1):273-89. doi: 10.1006/nimg.2001.0978. PMID 11771995
- [Background] Genovese CR, Lazar NA, Nichols T. Thresholding of statistical maps in functional neuroimaging using the false discovery rate. Neuroimage. 2002 Apr;15(4):870-8. doi: 10.1006/nimg.2001.1037. PMID 11906227
- [Background] Peltier SJ, Kerssens C, Hamann SB, Sebel PS, Byas-Smith M, Hu X. Functional connectivity changes with concentration of sevoflurane anesthesia. Neuroreport. 2005 Feb 28;16(3):285-8. doi: 10.1097/00001756-200502280-00017. PMID 15706237

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were screened out.
Groups:
- Initial MRI: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Anesthetics, Dissociative: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
Period: Overall Study
Arm/Group | Initial MRI | Hospital | Depresssion
Started | 3 | 7 | 3
Completed | 3 | 4 | 2
Not Completed | 0 | 3 | 1
Not completed — Researcher choice | 0 | 0 | 1
Not completed — Partial data analysis | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Initial Hospital; Depression: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
- Total: Total of all reporting groups
Arm/Group | Initial MRI | Initial Hospital | Depression | Total
Number analyzed (Participants) | 3 | 7 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 3 | 13
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 2 | 6 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Functional Connectivity
Description: The imaging experiments and analysis of subject-specific data will lead to maps corresponding to separate measures: resting state functional connectivity maps. The outcome of interest is whether ketamine reduces functional connectivity between the anterior (subgenual anterior cingulate corte, sgACC) and posterior regions (posterior cingulate cortex, PCC) of the default mode network. This is the z-score of the functional connectivity correlation.
  Timepoints for Initial fMRI were: Time 1:Immediately before Infusion, Time 2: After washout (Approx. 40 min after end of infusion).
  Timepoints for Depression were: Time 1: 1 Day before Infusion, Time 2: 1 Day after Infusion
Time Frame: 8 minutes scans, acquired between 1 day and 3 days (see above)
Population: Primary outcome measure is functional connectivity as measured using the MRI scans, which is only in the Initial MRI and Depression Arms.
Measure: Mean (Standard Error); unit: z score
Groups:
- Initial MRI: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
- Depression: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Anesthetics, Dissociative: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
Arm/Group | Initial MRI | Depression
Number analyzed (Participants) | 3 | 2
z score
  Before Infusion sgACC-PCC connectivity | 0.3114 (0.2199) | 0.3459 (0.018)
  After Infusion sgACC-PCC connectivity | -0.4424 (0.29) | 0.3208 (0.0465)

ADVERSE EVENTS:
Time Frame: Subjects were followed up for possible adverse events up to 4 weeks after the final infusion session.
Description: describe monitoring of subjects for adverse symptoms
Groups:
- Initial fMRI; Hospital; Depression: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
  Anesthetics, Dissociative: The subject will receive intravenous anesthesia at a dose of 0.5mg/kg delivered over 40 minutes in a constant infusion or bolus plus infusion method to maintain steady state (10 minutes initial induction, 30 minutes steady-state, for 40 minutes total)
Arm/Group | Initial fMRI | Hospital | Depression
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/7 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial fMRI (N=3) | Hospital (N=7) | Depression (N=3)
Discomfort (Psychiatric disorders) | 0 | 0 | 1 — One participant reported emotional discomfort with the dissociative effects of the intervention

LIMITATIONS AND CAVEATS:
These data should be interpreted with caution because of the small sample size due to the nature of this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No